# Telehealth CBT to address social isolation in Veterans with chronic pain

NCT05455476

April 2, 2024

# **Consent Script**

You are being invited to take part in this research because you have reported an impairment due to chronic pain and social isolation. This is a VA research study that hopes to learn more about how to address these issues. Our team has developed a non-medication intervention to help Veterans manage their pain and improve their mental health. This study will help us evaluate how well this treatment works.

# What is involved in the study?

Approximately 40 Veterans are expected to participate in this trial through the VA Finger Lakes Healthcare System to receive one of two types of treatment. Both treatments cover structured materials and exercises that involve strategies to manage pain, but one has more of an emphasis on feeling isolated from others. Using a procedure like the flip of a coin, participants will be randomly assigned to receive one of those two treatments. Both treatments consist of 8 weekly sessions that last approximately 45-60 minutes each.

If you decide to participate, you will be asked to complete some questionnaires about your pain and mental health that will take approximately 60-90 minutes to complete. These will occur by telehealth and will occur (1) prior to starting treatment (potentially today if you are available), (2) after treatment has been completed, (3) and about 30 days post-treatment completion.

Your interviews and your intervention sessions may be video and/or audio-recorded and if so, the recordings will be copied to a computer file on a secure VA computer server and then erased from the audio recorder as applicable. The recordings will be used to assure that the research staff is conducting the research study according to the study's protocol. The files will be deleted at the earliest opportunity consistent with applicable VA requirements. You are free to refuse to participate in this portion of the study and can still take part in the rest of the study.

# Confidentiality.

All the information collected will be treated as confidential. Electronic information will be kept on secure password-protected VA computers on servers behind the VA firewall. Any paper records will be kept in locked filing cabinets, within locked offices at the Center of Excellence for Suicide Prevention, which is a secure facility at the Canandaigua VA Medical Center. None of your identifying information will be connected to your responses. Your identifying information will not be connected to your responses, the information collected during this study, even if identifiers are removed, will not be used or distributed for future studies.

Importantly, none of this information will have any bearing on the healthcare that you receive. You proceed with your normal healthcare regardless of whether you choose to participate. At any time during this study, you can choose to withdraw from the study without prejudice or penalty. You can also choose not to answer any

question at any time without any bearing on the healthcare that you receive from the VA. Again, these research activities do not replace your care as usual. Therefore, if you are already engaged in treatment for pain or mental health, you will be encouraged to continue that treatment as appropriate and addressing ongoing concerns can be addressed with your regular treatment provider. If not engaged in care, but are interested in initiating treatment during or after the study, please let research staff know and we can provide a list of treatment resources for both within and outside the VA. If, however, you have any concerns about the ongoing study or your one time contact with our interventionist, you should feel free to bring that up with study staff or the primary investigator, Dr. Ashrafioun.

# What are the risks of participation?

Participation in this project is completely voluntary and you may withdraw at any time. Participation may involve risks that are unforeseeable. There is the possibility, though unlikely, that responding to questions on the survey may produce distress. Examples of distress include anxiety symptoms (e.g., shortness of breath, fear) or feeling down. If you experience distress during the interview, please discuss this with your interviewer. You may decide to stop the interview. If any significant new findings develop during the study that may affect your willingness to participate, we will provide you with this information in a timeline manner. We have no intention of sharing any of this information with your medical providers. However, if we are concerned about your safety, we will discuss it with you first and as a last resort reach out to emergency services if necessary. If you report any new medical concerns, we would encourage you to let your medical provider know of these concerns, but not contact them ourselves.

#### Are there benefits to participating in the study?

If you decide to take part in the study, there may or may not be direct medical benefits to you in terms of your mental health or medical conditions. However, you will be receiving treatment for your pain and mental health. We hope the information learned from the study will benefit other Veterans in the future as well. By conducting research studies such as this one, we can identify if this treatment can improve mental health outcomes and the management of pain.

You will receive compensation for your time for participating in the study. This compensation will be in the form of direct deposits, debit cards, or checks mailed to you by the VA following each completed session. The amount is as follows: Baseline assessment: \$40; Post-treatment assessment: \$40; 30-day follow-up: \$40.

The total compensation for completing all components of the study is \$120. Participants who do not complete the entire study for any reason will receive compensation for the components that were completed per the above pro-rated amounts and per the schedule of payments.

There is no cost to you for your participation.

If you have questions about this study or to report a research-related injury, you can contact: [redacted]. If you have general questions about giving your consent or your rights as a participant in this study or you would like to speak with an individual who is unaffiliated to this specific research study to discuss problems, concerns, and questions; obtain information or offer input you may call the Chairman of the Syracuse IRB or the Human Research Protection Program Administrator, at [redacted] or your local Patient advocate (https://www.va.gov/health/patientadvocate/).

At the final study appointment, we may ask if you're interested in other related studies. Whether or not you are interested, we will not retain your information for future contact unless you ask us directly to contact you at another time about any other opportunities. When applicable, this information will be kept behind a secure VA firewall and will only be accessible to approved study staff.

Do you have any questions? Would you like to participate in the study today?

\*If the individual agrees to participate in the study, proceed with the Comprehension of Verbal Informed

Consent below\*

# **Comprehension of Verbal Informed Consent**